CLINICAL TRIAL: NCT01889693
Title: Identification of Vascular Inflammatory Image Using a 68Ga-MSA(Gallium-68 Neomannosyl Human Serum Albumin) in Patients With Atherosclerotic Lesions
Brief Title: Imaging of Atherosclerosis With 68Ga-MSA
Status: Completed | Type: Observational
Sponsor: Korea University (Other)
Collaborators: Ministry of Health & Welfare, Korea (Other Government)
Responsible Party: Principal Investigator, Hong Seog Seo, Professor of Medicine, Korea University
Other Study IDs: GaMSA-Atherosclerosis
Record Dates: First submitted 2013-06-26; First posted 2013-06-28 (Estimated); Last update posted 2013-08-27 (Estimated); Status verified 2013-08

CONDITIONS: Atherosclerosis; Noninvasive Imaging of Atherosclerosis
Keywords: positron emission tomography; macrophage; neomannosyl human serum albumin
MeSH Terms: conditions — Atherosclerosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- acute coronary syndrome: patients with acute myocardial infarction and unstable angina
- chronic stable angina: patients with chronic stable angina
- control: control subjects without coronary artery disease

SUMMARY:
Despite of intensive efforts, no specific ath¬erosclerosis-targeting agent labeled with positron emitter is not yet available. Fortunately, some scientists made the major advance in the field of clinical atherosclerosis molecular imaging by the metabolic PET reporter agent 18F(fluorine-18)-FDG(Fludeoxyglucose) applied to noninvasively image plaque macrophages in carotid arteries. However, coronary and cerebral arterial segments remain uninterpretable due to metabolic property of 18F-FDG. Applying the character of the terminal mannose residues of MSA binding with the mannose receptors of macrophages in atherosclerosis, we investigate whether 68Ga-MSA can be a novel agent for non-invasive molecular imaging of atherosclerotic lesion in PET.

ELIGIBILITY:
Inclusion Criteria:

* acute coronary syndrome(acute myocardial infarction, unstable angina)
* chronic stable angina
* control without coronary artery disease

Exclusion Criteria:

* pregnancy, allergy to albumin, chronic inflammatory disease

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: 20 patients with acute coronary syndrome, 20 patients with chronic stable angina and 20 control subjects wihout coronary artery disease of the Cardiovascular Center at Korea University Guro Hospital
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2012-08; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
comparison of SUV(standard uptake unit) at atherosclerotic plaque of aorta and carotid arteries among 3 groups | 1 day at the time of PET(positron emission tomogram) imaging

SECONDARY OUTCOMES:
side effect of PET imaging with 68Ga-MSA | with 7 days after PET imaging
  any side effects including changes of biochemical values and vital signs

CONTACTS AND LOCATIONS:
Locations (1):
- Korea University Guro Hospital, Seoul, South Korea